CLINICAL TRIAL: NCT03123913
Title: Study of Testosterone and rHGH in FSHD (STARFISH): A Proof-of-Concept Study
Brief Title: Study of Testosterone and rHGH in FSHD
Acronym: STARFISH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Chad Heatwole, Professor of Neurology, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R01NS095813-01 (NIH)
Record Dates: First submitted 2017-04-12; First posted 2017-04-21 (Actual); Results first posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Facioscapulohumeral Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral | interventions — testosterone enanthate; Testosterone Propionate; Human Growth Hormone; Growth Hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination therapy (Experimental): Testosterone Enanthate and Somatropin
  Interventions: Drug: Testosterone Enanthate; Drug: Somatropin

INTERVENTIONS:
Drug: Testosterone Enanthate — Testosterone enanthate in oil (140mg) delivered via intramuscular injections every 2 weeks.
  Other Names: Delatestryl; Tesostroval; Testro LA; Andro LA; Durathate; Everone; Testrin; Andropository; Testosterone heptanoate
Drug: Somatropin — Genotropin (5.0 μg/kg/day) delivered via subcutaneous injections.
  Other Names: Genotropin; Humatrope; Norditropin; Nutropin; Serostim; Zorbtive

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of combination therapy with recombinant human growth hormone (rHGH) and testosterone in adult male patients with facioscapulohumeral muscular dystrophy (FSHD) over 24 weeks.

DETAILED DESCRIPTION:
This is a single-center, open-label study of daily human growth hormone (Genotropin®, 5.0 μg/kg via subcutaneous injection) and testosterone (testosterone enanthate, 140mg via intramuscular injection every two weeks) for 24 weeks in men with FSHD with a 12 week washout period. A total of 20 subjects will be enrolled at the University of Rochester Medical Center in Rochester, NY.

ELIGIBILITY:
Inclusion Criteria:

* A genetically confirmed diagnosis of FSHD (or clinical symptoms suggestive of FSHD with a first degree relative with genetically confirmed FSHD)
* Hematocrit of ≤ 50%
* Prostate-specific antigen ≤ 4.0 ng/ml (or ≤ 3.0 ng/ml if the participant has a first-degree relative with prostate cancer)
* Fasting blood glucose <126 mg/dl
* Able to walk continuously for six minutes (cane, walker, orthoses allowed)
* Able to independently administer intramuscular and subcutaneous injections (or have a family member who is capable and willing to administer these injections)

Exclusion Criteria:

* Diabetes
* Obesity (BMI>35 kg/m2)
* Cardiovascular disease (heart failure, coronary artery disease, uncontrolled hypertension, untreated hypercholesterolemia)
* Untreated thyroid disease
* Deep vein thrombosis
* Untreated severe sleep apnea
* Past pituitary disease
* Significant musculoskeletal injury and/or pain that affects walking
* A systolic blood pressure over 160 or a diastolic pressure over 100
* Plans to dramatically change exercise habits
* Liver disease
* Renal disease
* Cancer (other than basal cell skin cancer)
* Plans to conceive
* Heavy alcohol use (greater than 50g/day)
* Current testosterone or HGH use
* Current use of medications that interfere with the growth hormone or gonadal endocrine axis.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chad R Heatwole, MD, MS-CI, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Heatwole CR, Luebbe E, Hamel J, Mongiovi PC, Ciafaloni E, Dilek N, Martens WB, Weber DR, Rashid H, Allen McKeown J, Smith CH, Howell S, Rosero SZ, Eichinger K, Baker LS, Dekdebrun JM, Hilbert JE, Varma A, Thornton CA, McDermott MP, Moxley RT 3rd. Study of Testosterone and Recombinant Human Growth Hormone in Facioscapulohumeral Muscular Dystrophy. Neurol Genet. 2025 Aug 27;11(5):e200292. doi: 10.1212/NXG.0000000000200292. eCollection 2025 Oct. PMID 40900971

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination Therapy
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Combination Therapy
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an AE
Description: AEs were collected through patient report, interval laboratory studies, resting echocardiograms, dual energy x-ray absorptiometry (DEXA) studies, and physical examinations.
Time Frame: 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 20
Participants | 14

2. Secondary Outcome: Mean Change in Level of Free Testosterone in the Blood
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Combination Therapy
Number analyzed (Participants) | 19
pg/mL | 17.42 (77.94)

3. Secondary Outcome: Mean Change in Level of Total Testosterone in the Blood
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Combination Therapy
Number analyzed (Participants) | 19
ng/dL | 8.26 (277.94)

4. Secondary Outcome: Mean Change in Level of IGF-1 in the Blood
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Combination Therapy
Number analyzed (Participants) | 19
ng/mL | 89.79 (71.57)

5. Secondary Outcome: Mean Change in Level of TSH in the Blood
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Combination Therapy
Number analyzed (Participants) | 19
uIU/mL | 0.37 (0.66)

6. Secondary Outcome: Mean Change in Level of Luteinizing Hormone in the Blood
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Combination Therapy
Number analyzed (Participants) | 19
mIU/mL | -3.48 (2.64)

7. Secondary Outcome: Mean Change in Level of FSH in the Blood
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Combination Therapy
Number analyzed (Participants) | 19
mIU/mL | -3.29 (4.47)

8. Secondary Outcome: Mean Change in Total Lean Body Mass
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Combination Therapy
Number analyzed (Participants) | 19
Kg | 2.21 (1.79)

ADVERSE EVENTS:
Time Frame: 36 weeks
Arm/Group | Combination Therapy
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy (N=20)
Decreased energy (General disorders) | 1
Exercise fatigue (General disorders) | 1
Soreness (General disorders) | 2
Increased appetite (General disorders) | 2
Itchiness (General disorders) | 1
Poison ivy (Skin and subcutaneous tissue disorders) | 1
Vivid dreams (Psychiatric disorders) | 1
Elevated IGF-1 (Blood and lymphatic system disorders) | 3
Elevated testosterone (Blood and lymphatic system disorders) | 1
Elevated HbA1c (Blood and lymphatic system disorders) | 1
Elevated insulin (Blood and lymphatic system disorders) | 1
Elevated HCT (Blood and lymphatic system disorders) | 1
Elevated glucose (Blood and lymphatic system disorders) | 1
Glycosuria (Renal and urinary disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Parathesia (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Edema limbs (General disorders) | 2
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 1
Flu-like symptoms (General disorders) | 2
Headache (Nervous system disorders) | 1
Injection site reaction (General disorders) | 7
Irritability (Psychiatric disorders) | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pain (General disorders) | 2
Palpitations (Cardiac disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Urine discoloration (Renal and urinary disorders) | 1
Weight gain (Investigations) | 1
White patches on tongue (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT03123913/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT03123913/ICF_001.pdf